CLINICAL TRIAL: NCT03529487
Title: A Phase I, Open-Label, Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intra-anal Application of Topical Oxymetazoline Gel in Healthy Adult Volunteers
Brief Title: Intra-anal Oxymetazoline in Healthy Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RDD Pharma Ltd (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RDD 121
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Oxymetazoline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oxymetazoline applied intra analy (Experimental)
  Interventions: Drug: Oxymetazoline

INTERVENTIONS:
Drug: Oxymetazoline — Oxymetazoline gel applied intra-analy

SUMMARY:
This is a Phase 1, open-label, repeat dose, ascending dose study assessing the PK, safety, tolerability, PD, and dose- or exposure-response of Topical Oxymetazoline for intra-anal application. A total of 32 healthy male and female subjects will be enrolled to receive either Topical Oxymetazoline 1 mg (Cohort A, n=16), 5 mg (Cohort B, n=8) and 10 mg (Cohort C, n=8) applied intra-anally daily (QD) for 11 consecutive days.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, repeat dose, ascending dose study assessing the PK, safety, tolerability, PD, and dose- or exposure-response of Topical Oxymetazoline for intra-anal application.

The primary objective of this study is to determine the plasma concentrations and PK parameters, as data allows, of oxymetazoline following single and repeated intra-anal application of oxymetazoline gel 1 mg, 5 mg or 10 mg in healthy male and female subjects.

The secondary objective of this study is to evaluate the safety and tolerability of repeated intra-anal application of oxymetazoline gel 1 mg, 5 mg or 10 mg in healthy male and female subjects.

A total of 32 healthy male and female subjects will be enrolled (16 subjects in the first cohort and 8 subjects in the remaining cohorts) and will be exposed to Topical Oxymetazoline 1 mg, 5 mg or 10 mg applied intra-anally QD for 11 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
2. Subject is an adult male or female between the ages of 18 and 60 years, inclusive.
3. Female subjects of child-bearing potential must have a negative urine pregnancy test. Females of childbearing potential must practice a highly effective method of pregnancy prevention (defined as <1% pregnancies per 100 women per year) from one month before screening to one month after the follow-up visit, such as: surgical sterilization, hormonal implant, intrauterine device, or male condom + female diaphragm + vaginal spermicide. Female subject with any of the following circumstances is not required to use a highly effective method of pregnancy prevention: status post-hysterectomy; or, status post-tubal ligation; or, post-menopausal state (defined as >= 12 months of spontaneous amenorrhea) or < 12 months of spontaneous amenorrhea with a blood follicle stimulating hormone > 40 MIU/ml.
4. Subject has a body mass index between 18 and 33 kg/m2 (weight/[height]2).
5. Subject has normal (or abnormal and clinically insignificant) laboratory values at Screening.
6. Subject is healthy based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring and have no more than 3 spontaneous bowel movements (SBM) a day or no less than 3 SBMs a week.
7. Based on single or averaged QTc values of triplicate ECGs over a brief recording period, QTc < 450 msec
8. Subject has the ability to understand the requirements of the study and a willingness to comply with all study procedures, including retaining a rectal gel for at least 60 min and undergoing repeat rectal manometries lasting 10-15 min.
9. Subject has not consumed and agrees to abstain from taking any prescription or non-prescription medications, including herbal and dietary supplements (such as St. John's wort) within 14 days prior to the first dose of study medication (except as authorized by the Investigator and Medical Monitor).
10. Subject has not consumed alcohol-containing beverages for 3 days prior to the first scheduled dose and agrees not to consume alcohol through the last study visit.
11. Subject has not used tobacco- and nicotine-containing products for 2 months prior to the first scheduled dose and agrees not to use through the last study visit.

Exclusion Criteria:

1. Subject has a hypersensitivity or allergy to oxymetazoline.
2. Subject has active or history of cardiovascular or cerebrovascular disease including hypertension, unstable angina, myocardial infarction, transient ischemic attacks/stroke, clinically significant arrhythmia, congestive heart failure, or cardiac valve abnormalities.
3. Subject has systolic blood pressure >130 mm Hg and/or diastolic blood pressure >80 mm Hg and/or resting heart rate >90 bpm or resting heart rate <50 bpm.
4. Subject has glaucoma (narrow-angle), Raynaud's disease/phenomenon, thromboangiitis obliterans, scleroderma, and/or Sjögren's syndrome.
5. Subject has diabetes per medical history or has fasting plasma glucose level > 7 mmol/l (126 mg/dl) at screening or has Glycated hemoglobin (HbA1C) ≥ 48 mmol/mol (≥ 6.5 DCCT %) at screening.
6. Subject has thyroid problems such as medical history of hypothyroidism, hyperthyroidism, sick euthyroid syndrome, thyroid cancer, thyroid surgery, Radioiodine treatment or enlarged thyroid upon physical examination, or thyroid nodule upon physical examination, or abnormal thyroid-stimulating hormone (TSH) at screening defined as level >4.0 mIU/mL or level <0.4 mIU/mL.
7. Subject with enlarged prostate as per medical history or per rectal examination in screening.
8. Subject has a history of rectal surgery.
9. Subject has upon physical examination a rectal deformation or signs of rectal disease such as fissure, hemorrhoids grade 3, rectal prolapse, fistula, infection or space occupying lesion.
10. Subjects with a history of or present symptoms related to irritable bowel disease, inflammatory bowel disease, or chronic constipation.
11. Subject reporting change in bowel habits in the last 14 days.
12. Subject reporting episodes of rectal bleeding in the last 90 days.
13. Subjects taking anticoagulants such as Coumarins, Heparins, and Factor Xa inhibitors.
14. Subjects taking drugs known to affect rectal tone: nitrates, calcium channel blockers, alpha antagonists, and alpha agonists.
15. Subjects taking beta-blockers, and/or cardiac glycosides.
16. Subjects taking anti-hypertensives such as diuretics, beta blockers, alpha antagonists, sympatholytics, ACE inhibitors, angiotensin II antagonists, renin inhibitors, calcium antagonists or direct vasodilators.
17. Subjects taking anti-diabetic medications such as insulin, Biguanides, α-Glucosidase Inhibitors, Dipeptidyl peptidase IV inhibitors, Insulin secretagogues, Sodium-glucose cotransporter 2 inhibitors, Thiazolidinediones, Amylin agonists, GLP-1 receptor-agonists.
18. Subjects taking drugs affecting the thyroid such as levothyroxine, propylthiouracil, methimazole or amiodarone.
19. Subject has a history illicit drug abuse in the past year or current evidence of such abuse in the opinion of the Investigator.
20. Subject has positive findings on urine drug/alcohol/cotinine screen.
21. Subject is positive for human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C on Screening assessments.
22. Subject has an abnormal screening lab results judged by the investigator as clinically significant.
23. Subject has thrombocytopenia defined as platelet level < 150,000 per microliter of blood.
24. Subject is pregnant or lactating.
25. Subject has an acute illness within 1 week of the first scheduled dose.
26. Subject has donated plasma within 7 days of drug administration.
27. Subject has donated 1 or more pints of blood (or equivalent blood loss) within 30 days prior to drug administration.
28. Subject has participated in an investigational drug study where the last assessment of that study was within the 30 days prior to the first scheduled dose of this study.
29. Subject is an immediate family member of personnel directly affiliated with the study, or is personally directly affiliated with the study at the investigative site, or is employed or related to the Sponsor, CRO or investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | 11 days
  Oxymetazoline Maximum observed plasma concentration
Tmax | 11 days
  Time to maximum concentration (Oxymetazoline), obtained directly from the observed concentration versus time data
AUClast | 11 days
  Oxymetazoline Area under the plasma concentration-time curve from time 0 to time of last measureable plasma concentration
t½ | 11 days
  Oxymetazoline Terminal elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States